CLINICAL TRIAL: NCT03367676
Title: 12 weekS Adjuvant dOcetaxel Plus trastuzumaB in Patients With Tumors ≤1cm, Node-negative, HER2-positive Breast cancER (SOBER):a Single-grouparm, Open-label, Prospective, Phase 2 Study
Brief Title: 12 weekS Adjuvant dOcetaxel Plus trastuzumaB in Patients With Small, Node-negative, HER2-positive Breast cancER (SOBER)
Acronym: SOBER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li Zhu, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1712
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: trastuzumab; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): 12 weeks adjuvant docetaxel plus trastuzumab
  Interventions: Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab is administered at a loading dose of 8 mg/kg IV followed by 6 mg/kg every 21 days for 4 cycles.
Drug: Docetaxel — Docetaxel 100mg/m2，d1，iv，q3w*4

SUMMARY:
This phase II trial aims to study the efficacy and safety of 12 weeks adjuvant docetaxel plus trastuzumab in patients with tumors ≤1cm, node-negative, HER2-positive breast cancer.

DETAILED DESCRIPTION:
Many clinical trials has showed the superiority of combining trastuzumab to chemotherapy in the treatment of HER2 positive early breast cancer with tumor size ≥1cm or node metastasis.But in pT1n0m0 breast cancer patients, patients with HER2 positive tumor show worse prognosis than those with HER2 negative tumor.A short duration of trastuzumab administration contaminately with chemotherapy may have similar efficacy and lowerer toxiticy compared with standard one year therapy.Our study aims to study the efficacy and safety of 12 weeks adjuvant docetaxel plus trastuzumab in patients with tumors ≤1cm, node-negative, HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Women aged ≥18 years

Have finished radical operation

Pathologically confirmed dignosis of infiltrating primary breast cancer

According to AJCC ,pT≤1cm, pN0,no evidence for metastasis

Operation specimens are available for ER, progesterone receptor (PR) and Her2 detection, patients should be Her2 positive tumor (3+ by IHC or FISH+ )

Has Eastern Cooperative Oncology Group (ECOG) Performance Score 0-1,expected survival time > 12 months

Adequate bone marrow function,adequate liver and renal function,and adequate coagulation function.

Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable and effective method of contraception to avoid pregnancy during the study.

Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

pT>1cm or node positive

Metastatic breast cancer

Any prior systemic or loco-regional treatment of breast cancer, including chemotherapy in 28 days

With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma

Patients with medical conditions that indicate intolerant to adjuvant chemotherapy and related treatment, including severe infection, coagulation disorder,active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease

Has symptomatic peripheral neuropathy > grade 2 according to NCI

Known severe allergy to any drugs in this study

Has cadiac Dysfunction or lung dysfunction defined as follows:

1. grade ≥3 CHF according to NCI CTCAE v 4.0 or NYHA≥II
2. angina which requires drug control ,cardiac infraction,and any other vascular disease with apparent clinical symptoms
3. uncontrolled high-risk arryhthmia
4. unconrolled hypertension

Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive

Patient is pregnant or breast feeding

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-12-30 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 3-year estimates
  Estimated percentage of patients alive and disease-free at 3 years from randomization, where disease-free survival is defined as the time from randomization to the first appearance of one of the following: invasive breast cancer recurrence at local, regional, or distant site, invasive contralateral breast cancer, second (non-breast) invasive cancer, or death without cancer event; or censored at date of last follow-up.

SECONDARY OUTCOMES:
Breast Cancer Specific Survival | 3-year estimates
  Estimated percentage of patients alive and disease-free at 3 years from randomization, where breast cancer specific survival is defined as the time from randomization to death from breast cancer relapse; or censored at date last known alive.
Overall Survival | 3-year estimats
  Estimated percentage of patients alive and disease-free at 3 years from randomization, where overall survival is defined as the time from randomization to death from any cause; or censored at date last known alive.
Treatment-related adverse events | up to 4 months
  Incidence and severity of adverse events as assessed by NCI CTCAE V4.0
Change of LVEF after treatment | up to 4 months
  The change of LVEF after 12 weeks treatment compared to the baseline LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhu, doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No